CLINICAL TRIAL: NCT01489176
Title: Regadenoson Stress Real-Time Myocardial Perfusion Echocardiography for Detection of Coronary Artery Disease Feasibility and Accuracy of Two Different Ultrasound Contrast Agents
Brief Title: Regadenoson Real Time Perfusion Imaging Trial-Optison
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Astellas Pharma US, Inc. (Industry); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0555-11-FB
Record Dates: First submitted 2011-12-02; First posted 2011-12-09 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Myocardial Perfusion Abnormalities
Keywords: Stress Echocardiography; Real-Time Perfusion Imaging; Regadenoson; Optison
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson; FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regadenoson; Optison (Experimental): Use of Regadenoson as the chemical stress agent using Optison as a contrast agent during stress echocardiography.
  Interventions: Drug: Regadenoson; Optison

INTERVENTIONS:
Drug: Regadenoson; Optison — A one-time intravenous bolus of Regadenoson 400 mcg; continuous intravenous infusion of Optison of 2-4 mL/minute.
  Other Names: Lexiscan is the brand name for regadenoson.

SUMMARY:
The purpose if this study is to examine how effective Regadenoson is in detecting coronary artery disease during a stress echocardiogram when Optison is administered. Optison is a contrast agent that improves the images of the heart on the echocardiogram (echo) machine. Optison is approved by the Food and Drug Administration (FDA) to use during stress echocardiograms. Regadenoson is a commercially available rapid acting stress agent that is used to chemically increase the heart rate and is approved for nuclear imaging tests. Regadenoson is a FDA approved drug but not for the intended use in this study.

DETAILED DESCRIPTION:
Stress perfusion imaging has primarily been done with radionuclide scintigraphy or single photon emission computed tomography (SPECT) and has not reached its full clinical potential because of the poor spatial resolution of SPECT, increased expense of this procedure, patient exposure to ionizing radiation, and lack of availability. The A2A receptor agonist Regadenoson has been utilized to detect myocardial perfusion abnormalities during SPECT myocardial perfusion imaging.

A 100 patient pilot study (Regadenoson Real Time Perfusion Imaging Trial, IRB #566-08-FB) demonstrated the feasibility and accuracy of real-time perfusion echocardiography (RTPE) in detecting coronary artery disease following Regadenoson bolus injection and Definity as an ultrasound contrast agent. The aim of this study is to determine whether similar feasibility and accuracy can be achieved with Optison (a Food and Drug Administration approved ultrasound contrast agent that differs slightly in microbubble size and composition) in detecting coronary artery disease (CAD) following Regadenoson bolus injection. As with the original study, sensitivity, specificity, and accuracy of perfusion and wall motion analysis to identify a coronary stenosis >50% in diameter by quantitative angiography will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female. Age ≥ 30 years.
* Resting Left Ventricular Ejection Fraction > 40% using Simpson's biplane measurement.
* Scheduled for coronary angiography within 30 days of the Regadenoson stress test.
* Negative urine pregnancy test within 2 hours of ultrasound contrast administration required of females of childbearing age unless post-menopausal or with evidence of surgical sterilization.
* Be conscious and coherent, and able to communicate effectively with trial personnel.
* Agreeable to undergo the additional stress test (which is being performed for research purposes only, not for clinical care) and coronary angiography (which is being performed for clinical care) based on the following clinical profile: Have at least an intermediate likelihood of coronary disease based.
* Good apical echo images with at least 50% of each coronary artery territory well visualized.

Exclusion Criteria:

* Known or suspected hypersensitivity to ultrasound contrast agent used for the study.
* Pregnancy or lactation.
* Complicated hemodynamic instability (i.e., NYHA Class IV heart failure, unstable angina at rest despite medical therapy).
* Life expectancy of less than two months or terminally ill.
* Congestive (idiopathic) or hypertrophic cardiomyopathy.
* Known left main disease.
* Heart transplant recipient, hypertrophic cardiomyopathy, acute myo- or pericarditis.
* Resting Left Ventricular Ejection Fraction < 40%
* Large inducible perfusion defects or wall motion abnormalities during prior stress imaging study associated with left ventricular cavity dilatation.
* Early positive treadmill ECG within the first stage of the test.
* History of > 1st degree heart block, sick sinus syndrome or high grade AV block without a pacemaker.
* Dipyridamole use within 30 hours of stress test, or consumption of methylxanthines within 12 hours, or use of sublingual nitroglycerin within two hours.
* Participation in another investigational study within one month of this study.
* Anyone in whom a stress test should not be performed prior to cardiac catheterization.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- See also: Journal of the American Society of Echocardiography — https://doi.org/10.1016/j.echo.2015.08.011

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regadenoson; Optison
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regadenoson; Optison
Number analyzed (Participants) | 50
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 62 [51 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 50
BMI [Mean (Inter-Quartile Range); unit: kg/m2] | 32 [25 to 39]
Percutaneous coronary intervention (PCI) Coronary artery bypass surgery (CABG) [Count of Participants; unit: Participants] — Percutaneous coronary intervention (PCI) Coronary artery bypass surgery (CABG)
  Participants | 17
Hypertension [Number; unit: participants] | 40
Hyperlipidemia [Number; unit: participants] | 47
Diabetes [Count of Participants; unit: Participants] | 17
Resting ejection fraciton (%) [Log Mean (Inter-Quartile Range); unit: percent] | 57 [50 to 65]
Resting heart rate, bpm [Mean (Full Range); unit: beats per minute] | 67 [55 to 79]
Peak heart rate, bpm [Mean (Inter-Quartile Range); unit: beats per minute] | 84 [72 to 96]
Resting SBP, mm Hg [Mean (Inter-Quartile Range); unit: mm Hg] | 130 [108 to 152]
Peak SBP, mm Hg [Mean (Inter-Quartile Range); unit: mm Hg] | 124 [103 to 145]
Resting DBP, mm Hg [Mean (Inter-Quartile Range); unit: mm Hg] | 73 [60 to 86]
Peak Diastolic Blood Pressure (DBP) [Mean (Inter-Quartile Range); unit: mm Hg] | 67 [58 to 76]
Resting Rate Pressure Product (RPP) [Mean (Standard Deviation); unit: beats/minute*mmHg] | 8754 (1846)
Peak Rate Pressure Product (RPP) [Mean (Standard Deviation); unit: beats/minute*mmHg] | 11,738 (2,862)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Coronary Stenosis
Description: Measurements will be analyzed to identify a coronary stenosis >50% in diameter by quantitative cardiac angiography.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Regadenoson; Optison
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Arm/Group | Regadenoson; Optison
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 50/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regadenoson; Optison (N=50)
Chest Pain (Cardiac disorders) | 7 (7)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 26 (26)
Headaches (General disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No